CLINICAL TRIAL: NCT00731731
Title: Phase I/II Study of Vorinostat (Suberoylanilide Hydroxamic Acid [SAHA]), Temozolomide, and Radiation Therapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: Vorinostat, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00672; NCI-2009-00672 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N0874; ABTC 0902; CDR0000609743; N0874 (Other: Alliance for Clinical Trials in Oncology); N0874 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; Mental Status and Dementia Tests; Temozolomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy, vorinostat, temozolomide) (Experimental): Patients undergo radiotherapy and receive vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive vorinostat PO QD on days 1-7 and 15-21 and temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Cognitive Assessment; Other: Laboratory Biomarker Analysis; Drug: Temozolomide; Drug: Vorinostat

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Procedure: Cognitive Assessment — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I/II trial studies the side effects and best dose of vorinostat when given together with temozolomide and radiation therapy and to see how well they work in treating patients with newly diagnosed glioblastoma multiforme. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving vorinostat together with temozolomide and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of vorinostat in patients with newly diagnosed glioblastoma multiforme (GBM) and gliosarcomas, who are also receiving concomitant radiation therapy (RT) and temozolomide (TMZ). (Phase I) II. To define the safety of vorinostat with RT and TMZ in this population. (Phase II) III. To determine the efficacy of vorinostat in combination with RT and TMZ followed by vorinostat in combination with TMZ in patients with newly-diagnosed GBM and gliosarcomas as measured by overall survival at 15 months (OS15). (Phase II)

SECONDARY OBJECTIVES:

I. To determine progression-free survival in newly diagnosed GBM and gliosarcoma patients treated with the study regimen. (Phase II) II. To further evaluate the safety profile of vorinostat in combination with RT and TMZ in this patient population. (Phase II) III. Determine the neurocognitive effects in patients treated on this protocol and correlate these results with outcome endpoints. (Phase II)

TERTIARY OBJECTIVES:

I. To explore the extent to which the tumor's molecular characteristics and expression profile correlate with outcome.

II. Evaluate potential mechanisms of therapy resistance in tumor samples obtained at the time of tumor progression.

OUTLINE: This is a phase I, dose-escalation study of vorinostat followed by a phase II study.

Patients undergo radiotherapy and receive vorinostat orally (PO) once daily (QD) on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive vorinostat PO QD on days 1-7 and 15-21 and temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 1 year, every 3 months for 1 year and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION:
* Central pathology review submission; this review is mandatory prior to registration to confirm eligibility; it should be initiated as soon after surgery as possible
* Treatment should begin >= 2 weeks and =< 5 weeks following surgery
* REGISTRATION:
* Histologically confirmed glioblastoma multiforme as determined by pre-registration central pathology review; Note: gliosarcomas and other grade 4 astrocytoma variants (e.g., giant cell) are eligible
* Measurable or evaluable disease by gadolinium magnetic resonance imaging (MRI) or contrast computed tomography (CT) scan; Note: patients who have had a gross total resection (GTR) are eligible on the basis of evaluable disease

  * Must begin partial brain radiotherapy on the same day that vorinostat and temozolomide begin
* Karnofsky performance status of >= 60
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* White blood cell (WBC) >= 3,000/mm^3
* Hemoglobin >= 10.0 g/dL; Note: this level may be reached by transfusion
* Total bilirubin =< 2.0 x institutional upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.0 x ULN
* Creatinine =< 1.5 mg/dL
* Life expectancy >= 12 weeks
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* For Phase I established MTD and Phase II patients only: Willing and able to complete neurocognitive testing
* Ability to provide informed written consent
* Willing to return to Alliance or Adult Brain Tumor Consortium (ABTC) enrolling institution for follow-up
* Phase I established MTD patients and Phase II patients: Willing to provide mandatory tissue samples (slides or blocks) for research purposes
* Willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while being treated with vorinostat and temozolomide

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the duration of the study and for 12 weeks after treatment has ended
* Prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors
* Prior cranial RT
* Prior Gliadel wafers
* Known hypersensitivity to any of the components of vorinostat or other agents used in study
* Valproic acid, another histone deacetylase inhibitor, =< 2 weeks prior to registration and during treatment
* Other active malignancy =< 3 years prior to registration; Exception: non-melanotic skin cancer or carcinoma in situ of the cervix; Note: if there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* Uncontrolled infection
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; Note: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Co-morbid systemic illness or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with proper assessment of safety and adverse events of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* History of myocardial infarction or unstable angina =< 6 months prior to registration or congestive heart failure (CHF) requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* New York Heart Association (NYHA) >= Class II Congestive Heart Failure
* Inability to take oral medications
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Congenital long QT syndrome
* Prolonged corrected (QTc) interval (> 450 msec)
* Any of the following Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes =< 7 days prior to registration

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-07-10 (Actual); Primary Completion 2014-02-02 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (110):
- United States (110):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Cancer Trials Support Unit, Rockville, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin

REFERENCES:
- [Derived] Cerhan JH, Anderson SK, Butts AM, Porter AB, Jaeckle K, Galanis E, Brown PD. Examiner accuracy in cognitive testing in multisite brain-tumor clinical trials: an analysis from the Alliance for Clinical Trials in Oncology. Neurooncol Pract. 2019 Jul;6(4):283-288. doi: 10.1093/nop/npy048. Epub 2018 Nov 24. PMID 31386061

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose Level 0: Patients undergo 60 Gy radiotherapy and receive 300 mg vorinostat PO QD (every day) on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 500 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * dimensional conformal radiation therapy: Undergo radiotherapy > > temozolomide: Given PO > > vorinostat: Given PO > > cognitive assessment: Ancillary studies > > laboratory biomarker analysis: Correlative studies
- Phase I, Dose Level 1: Patients undergo 60 Gy radiotherapy and receive 400 mg vorinostat PO QD (every day) on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 500 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * dimensional conformal radiation therapy: Undergo radiotherapy > > temozolomide: Given PO > > vorinostat: Given PO > > cognitive assessment: Ancillary studies > > laboratory biomarker analysis: Correlative studies
- Phase II: Patients undergo 60 Gy radiotherapy and receive 300 mg vorinostat PO QD (every day) on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 400 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5 for cycle 2 and 200 mg/m2 temozolomide PO QD on days 1-5 for all subsequent cycles. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * dimensional conformal radiation therapy: Undergo radiotherapy > > temozolomide: Given PO > > vorinostat: Given PO > > cognitive assessment: Ancillary studies > > laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase II
Started | 12 | 3 | 110
Completed | 12 | 3 | 107
Not Completed | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Cancel prior to treatment | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase I, Dose Level 0: Patients undergo 60 Gy radiotherapy and receive 300 mg vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 500 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  * dimensional conformal radiation therapy: Undergo radiotherapy> > temozolomide: Given PO> > vorinostat: Given PO> > cognitive assessment: Ancillary studies> > laboratory biomarker analysis: Correlative studies
- Phase I, Dose Level 1: Patients undergo 60 Gy radiotherapy and receive 400 mg vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 500 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  * dimensional conformal radiation therapy: Undergo radiotherapy> > temozolomide: Given PO> > vorinostat: Given PO> > cognitive assessment: Ancillary studies> > laboratory biomarker analysis: Correlative studies
- Phase II: Patients undergo 60 Gy radiotherapy and receive 300 mg vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 400 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5 for cycle 2 and 200 mg/m2 temozolomide PO QD on days 1-5 for all subsequent cycles. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  * dimensional conformal radiation therapy: Undergo radiotherapy> > temozolomide: Given PO> > vorinostat: Given PO> > cognitive assessment: Ancillary studies> > laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase II | Total
Number analyzed (Participants) | 12 | 3 | 107 | 122
Age, Continuous [Median (Full Range); unit: years] | 57 [43 to 76] | 59 [58 to 73] | 59 [20 to 80] | 59 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 44 | 51
  Male | 8 | 0 | 63 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 4
  White | 12 | 3 | 99 | 114
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Vorinostat, Defined as the Dose at Which Fewer Than One-third of Patients Experience DLTs, Graded According to NCI CTCAE (Common Toxicity Criteria for Adverse Effects) Version 3.0 (Phase I)
Description: The Maximum Tolerated Dose (MTD) will be based on the assessment of Dose Limiting Toxicity (DLT) during the first 10 weeks of treatment only, and will be defined as the dose at which fewer than one-third of patients experience a DLT to vorinostat. The MTD is the dose level at which 0/3 or 1/6 patients experience DLT with the next higher dose having at least 2/3 or 2/6 patients encountering DLT.
  >
  >
  DLT will be defined as any of the following events occurring during treatment with vorinostat and temozolomide and attributable to one or both study drugs:
  * Grade 3 or 4 thrombocytopenia, grade 4 anemia or grade 4 neutropenia lasting > 7 days
  * Any non-hematologic grade 3 or greater adverse event, excluding alopecia and venous thromboembolism
  * Grade 4 radiation-induced skin changes
  * Failure to recover from toxicities to be eligible for re-treatment with vorinostat and temozolomide ≤ 14 days of the last dose of the two drugs
Time Frame: 10 weeks
Measure: Number; unit: number of patients with DLT
Groups:
- Phase I, Dose Level 0: Patients undergo 60 Gy radiotherapy and receive 300 mg vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 500 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * dimensional conformal radiation therapy: Undergo radiotherapy > > temozolomide: Given PO > > vorinostat: Given PO > > cognitive assessment: Ancillary studies > > laboratory biomarker analysis: Correlative studies
- Phase I, Dose Level 1: Patients undergo 60 Gy radiotherapy and receive 400 mg vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 500 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * dimensional conformal radiation therapy: Undergo radiotherapy > > temozolomide: Given PO > > vorinostat: Given PO > > cognitive assessment: Ancillary studies > > laboratory biomarker analysis: Correlative studies
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1
Number analyzed (Participants) | 12 | 3
number of patients with DLT | 3 | 3

2. Primary Outcome: Overall Survival at 15 Months (Phase II)
Description: The primary endpoint will be survival status at 15 months (OS15). In addition, survival will be estimated using a Kaplan-Meier curve. For this analysis, patients who are still alive at the time of analysis have survival time censored at the last contact date.
Time Frame: Time from study registration to the date of death from any cause, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of phase II patients
Groups:
- Phase II: Patients undergo 60 Gy radiotherapy and receive 300 mg vorinostat PO QD on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients also receive 75 mg/m2 temozolomide PO QD on days 1-42. Beginning 4-6 weeks later, patients receive 400 mg vorinostat PO QD on days 1-7 and 15-21 and 150 mg/m2 temozolomide PO QD on days 1-5 for cycle 2 and 200 mg/m2 temozolomide PO QD on days 1-5 for all subsequent cycles. Treatment with vorinostat and temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  * dimensional conformal radiation therapy: Undergo radiotherapy > > temozolomide: Given PO > > vorinostat: Given PO > > cognitive assessment: Ancillary studies > > laboratory biomarker analysis: Correlative studies
Arm/Group | Phase II
Number analyzed (Participants) | 107
percentage of phase II patients | 54.6 [45.9 to 65.0]

3. Secondary Outcome: Incidence of Adverse Events, Based on CTC (Common Toxicity Criteria) Severity Grade
Description: Safety variables will be summarized by descriptive statistics. Adverse Events (AEs) that occur will be reported for each phase and dose level and described in terms of incidence and severity. Parameters will be described based on the CTC severity grading. Distribution by CTC severity grade and clinical relevance will be given.
Time Frame: Up to 5 years
Measure: Number; unit: participants evaluable for toxicity
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase II
Number analyzed (Participants) | 12 | 3 | 107
participants evaluable for toxicity | 12 | 3 | 107

4. Secondary Outcome: Time to Tumor Progression (Phase II)
Description: Progression free survival time will be defined from date of registration to date of progression or death.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 107
months | 8.05 [6.21 to 9.30]

5. Secondary Outcome: Incidence of Adverse Events, as Per NCI CTCAE Version 3.0 (Phase II)
Description: The maximum grade for each type of treatment-related adverse event will be recorded for each patient, and frequency tables for each arm will be reviewed to determine patterns. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing.
Time Frame: Up to 5 years
Measure: Number; unit: participants evaluable for toxicity
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase II
Number analyzed (Participants) | 12 | 3 | 107
participants evaluable for toxicity | 12 | 3 | 107

ADVERSE EVENTS:
Groups:
- Phase I, Dose Level 0; Phase I, Dose Level 1; Phase II: laboratory biomarker analysis: Correlative studies
Arm/Group | Phase I, Dose Level 0 | Phase I, Dose Level 1 | Phase II
Serious Adverse Events (participants affected / at risk) | 11/12 | 1/3 | 63/107
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 106/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 0 (N=12) | Phase I, Dose Level 1 (N=3) | Phase II (N=107)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 11 (26)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (3)
Fatigue (General disorders) | 0 (0) | 1 (1) | 10 (17)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
General symptom (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 8 (13)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (6)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 1 (1) | 19 (54)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4) | 0 (0) | 18 (61)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 17 (47)
Platelet count decreased (Investigations) | 4 (4) | 1 (1) | 25 (81)
Weight loss (Investigations) | 0 (0) | 0 (0) | 3 (11)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (14)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (11)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (8)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 16 (39)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 0 (N=12) | Phase I, Dose Level 1 (N=3) | Phase II (N=107)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (28) | 1 (1) | 91 (704)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (7)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (16)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 4 (5)
Flashing vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 7 (22)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 3 (16)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 13 (28)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 40 (171)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 0 (0) | 37 (119)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (34)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (24)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (6)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (13)
Nausea (Gastrointestinal disorders) | 6 (25) | 1 (1) | 70 (386)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (10) | 1 (1) | 38 (92)
Chills (General disorders) | 0 (0) | 0 (0) | 5 (6)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 7 (13)
Fatigue (General disorders) | 12 (53) | 2 (2) | 103 (942)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 8 (36)
Localized edema (General disorders) | 0 (0) | 0 (0) | 2 (4)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (7)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (5)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 9 (19)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (10)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 31 (69)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 25 (53)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 13 (51)
Creatinine increased (Investigations) | 3 (12) | 0 (0) | 14 (56)
INR increased (Investigations) | 0 (0) | 1 (1) | 1 (4)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Leukocyte count decreased (Investigations) | 9 (30) | 0 (0) | 65 (358)
Lymphocyte count decreased (Investigations) | 7 (27) | 2 (2) | 51 (256)
Neutrophil count decreased (Investigations) | 6 (14) | 0 (0) | 50 (198)
Platelet count decreased (Investigations) | 8 (44) | 2 (2) | 91 (584)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight gain (Investigations) | 0 (0) | 0 (0) | 3 (8)
Weight loss (Investigations) | 1 (1) | 0 (0) | 17 (53)
Anorexia (Metabolism and nutrition disorders) | 5 (17) | 2 (2) | 62 (274)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (3) | 3 (3) | 14 (41)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 23 (32)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (9)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 12 (20)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (8)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 9 (15)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 14 (26)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 13 (25)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 9 (17)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (25)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (30)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (12)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (19)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (6)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 4 (16)
Cognitive disturbance (Nervous system disorders) | 4 (11) | 0 (0) | 35 (194)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 7 (28)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 24 (86)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 6 (14) | 1 (1) | 44 (289)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 5 (33)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 7 (27)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 8 (28)
Taste alteration (Nervous system disorders) | 6 (24) | 1 (1) | 53 (283)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 8 (20)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (6)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (9)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 8 (19)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 17 (46)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (5)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (11)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 9 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (15)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (8) | 0 (0) | 33 (138)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (10)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (16)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (8)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (6)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 5 (29)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less